CLINICAL TRIAL: NCT00087217
Title: Phase I Study of 17- Allylamino-17 Demethoxygeldanamycin (17-AAG) in Combination With Paclitaxel in Advanced Solid Malignancies
Brief Title: 17-N-Allylamino-17-Demethoxygeldanamycin and Paclitaxel in Treating Patients With Metastatic or Unresectable Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02610; PCI-03-152; U01CA099168 (NIH); U01CA062502 (NIH); CDR0000373824 (Registry Identifier: PDQ (Physician data Query))
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — tanespimycin; Paclitaxel; Taxes

ARMS (1):
- Treatment (tanespimycin, paclitaxel) (Experimental): Patients receive 17-AAG IV over 1 hour on days 1*, 4, 8, 11, 15 and 18 and paclitaxel IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tanespimycin; Drug: paclitaxel; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of 17-N-allylamino-17-demethoxygeldanamycin when given together with paclitaxel in treating patients with metastatic or unresectable solid tumor. Drugs used in chemotherapy, such as 17-N-allylamino-17-demethoxygeldanamycin and paclitaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining 17-N-allylamino-17-demethoxygeldanamycin with paclitaxel may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) when administered with paclitaxel in patients with metastatic or unresectable solid malignancy.

II. Determine the dose-limiting and non-dose-limiting toxic effects of this regimen in these patients.

III. Determine the pharmacokinetics of this regimen in these patients. IV. Determine tumor response in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG). Patients receive 17-AAG IV over 1 hour on days 1*, 4, 8, 11, 15 and 18 and paclitaxel IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *17-AAG is not administered on day 1 of course 1. Cohorts of 3-6 patients receive escalating doses of 17-AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 6-12 patients are treated at the recommended phase II dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid malignancy

  * Metastatic or unresectable disease
* Not amenable to standard curative or palliative therapy
* No known brain metastases
* Performance status - ECOG 0-2
* More than 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3
* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin normal
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* QTc < 450 msec for male patients (470 msec for female patients)
* LVEF > 40% by MUGA
* No history of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No myocardial infarction within the past year
* No New York Heart Association class III or IV congestive heart failure
* No poorly controlled angina
* No history of uncontrolled dysrhythmia or requirement for antiarrhythmic drugs
* No history of congenital long QT syndrome
* No active ischemic heart disease within the past year
* No left bundle branch block
* No other significant cardiac disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double barrier contraception for at least 1 week before, during, and for at least 2 weeks after study participation
* No prior allergy to eggs
* No prior allergic reaction to compounds of similar chemical or biologic composition to 17-AAG or paclitaxel
* No peripheral neuropathy > grade 1
* No concurrent uncontrolled illness
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* No concurrent granulocyte colony-stimulating factors
* Prior paclitaxel allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior 17-N-allylamino-17-demethoxygeldanamycin (17-AAG)
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy that included the heart in the field (e.g., mantle radiotherapy)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent therapeutic-dose warfarin for anticoagulation
* No concurrent medications that may prolong QTc interval
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-05; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Phase 2 recommended doses of tanespimycin | 28 days
  Tabulated according to the NCI CTC.

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Ramalingam, Principal Investigator — University of Pennsylvania Medical Center
Locations (1):
- University of Pennsylvania Medical Center, Philadelphia, Pennsylvania, United States